CLINICAL TRIAL: NCT04010383
Title: Non-inferiority Study for Visual Field Measurements Using a Virtual Reality Device on Participants With Normal and Glaucomatous Visual Fields
Brief Title: Non-inferiority Study for Visual Field Measurements Using a Virtual Reality Device
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01902
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Visual Field Tests
Keywords: Perimetry; Virtual reality device

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal visual field subjects: * Cataract yes or no
  * Age range 40 - 80 years
  * normal visual field (MD: < +2 dB)
  * Refractive error within ±5 dpt. spherical equivalent
  * Astigmatism of < -3 dpt.
  * Visual acuity of ≥0.3 logMar (decimal ≥0.5)
  * Experience in perimetry (history of at least one perimetry examination)
  * False positive or negative errors each less than 20% in each examination
  Interventions: Diagnostic Test: virtual reality perimeter
- Glaucomatous subjects: * Primary open-angle/ pseudoexfoliation/ primary angle-closure glaucoma
  * Early to moderate visual field loss (MD: +2 to +12 dB)
  * Refractive error within ±5 dpt. spherical equivalent
  * Astigmatism of < -3 dpt.
  * Visual acuity of ≥0.3 logMar (decimal ≥0.5)
  * Experience in perimetry (history of at least one perimetry examination)
  * False positive or negative errors each less than 20% in each examination
  * Cataract yes or no
  * Age range 40 - 80 years
  Interventions: Diagnostic Test: virtual reality perimeter

INTERVENTIONS:
Diagnostic Test: virtual reality perimeter — Both groups will be examined with a standard automated perimeter as well as with the virtual reality perimeter.

SUMMARY:
It is hypothesized that performing VF measurements with a Virtual Reality headset using similar testing strategies as implemented in conventional perimeters, allow for a non-inferior quality in VF acquisitions. The results of this study will show if valid measurements of such devices in human subjects can be obtained.

The primary endpoint of this study is the non-inferiority estimation quality of participant's mean defect (MD) measured in decibel (dB) between the head-mounted display and an OCTOPUS perimeter using the dynamic strategy (DS) for participants with normal or glaucomatous visual field. The MD is a clinical measure for the average loss of visual function calculated from the visual field of a participant.

ELIGIBILITY:
Written informed consent

Inclusion Criteria for normal visual field subjects:

* Cataract yes or no
* Age range 40 - 80 years- normal visual field (MD: < +2 dB)
* Refractive error within ±5 dpt. spherical equivalent
* Astigmatism of < -3 dpt.
* Visual acuity of ≥0.3 logMar (decimal ≥0.5)
* Experience in perimetry (history of at least one perimetry examination)
* False positive or negative errors each less than 20% in each examination

Inclusion Criteria for glaucomatous subjects:

* Primary open-angle/ pseudoexfoliation/ primary angle-closure glaucoma
* Early to moderate visual field loss (MD: +2 to +12 dB)
* Refractive error within ±5 dpt. spherical equivalent
* Astigmatism of < -3 dpt.
* Visual acuity of ≥0.3 logMar (decimal ≥0.5)
* Experience in perimetry (history of at least one perimetry examination)
* False positive or negative errors each less than 20% in each examination
* Cataract yes or no

Exclusion Criteria:

* Exclusion criteria are subjects younger than 40 and older than 80 years
* Inability to follow the procedure
* Insufficient knowledge of project language
* The history of other ocular diseases than glaucoma or cataract or other conditions that might affect visual field testing (e.g. pituitary lesions, demyelinating diseases).
* Any history of epilepsy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of glaucoma patients and patients with normal visual fields respecting the inclusion/exclusion criteria. There is no restriction in ethnicity.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
non-inferiority estimation quality of mean defect (MD) measured in decibels (dB) between the virtual reality perimeter and the OCTOPUS 900 perimeter | 2 weeks
  The primary endpoint of this study is the non-inferiority estimation quality of participant's mean defect (MD) measured in decibel (dB) between the head-mounted display and an OCTOPUS perimeter using the dynamic strategy (DS) for participants with normal or glaucomatous visual field. The MD is a clinical measure for the average loss of visual function calculated from the visual field of a participant.

CONTACTS AND LOCATIONS:
Overall Officials: René G Höhn, Dr. med., Principal Investigator — Department of Ophthalmology, University Hospital Bern, Berne, Switzerland
Locations (1):
- University Hospital Bern, Department of Ophthalmology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No